CLINICAL TRIAL: NCT04689061
Title: A Multi-Center, Prospective Study to Evaluate the Continued Safety and Effectiveness of the FastThread Interference Screws
Brief Title: FastThread Interference Screws
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arthrex, Inc. (Industry)
Collaborators: Arthrex GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0011
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Biocomposite FastThread Interference Screw: The absorbable Biocomposite Interference Screws combine the inherent degradation characteristics of a biocompatible polymer with the bioactivity of a ceramic. They are made of a combination of 70% poly (L-lactide-co-D, L-lactide) (PLDLA) and 30% biphasic calcium phosphate (BCP). The material has withstood the test of time with over a decade of clinical use and millions of implantations. It has been shown that the Biocomposite Interference Screw integrates well into the surrounding bone, produces little to no inflammatory response, and partially degrades 2 years after implantation
  Interventions: Device: Arthrex FastThread Interference Screw

INTERVENTIONS:
Device: Arthrex FastThread Interference Screw — The Arthrex PEEK and Biocomposite FastThread Interference Screws have a tapered hexalobe design along the entire length of the screw to maximize transfer of torque and reduce screw stripping. The Arthrex PEEK and Biocomposite FastThread Interference Screws have a tapered hexalobe design along the entire length of the screw to maximize transfer of torque and reduce screw stripping

SUMMARY:
Surgery using the Arthrex PEEK or Biocomposite FastThread Interference Screw for ACL or PCL (PCL at US sites only, Biocomposite screw PCL only) repair or reconstruction.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the continued safety and effectiveness of the PEEK and Biocomposite FastThread Interference Screws used for Anterior Cruciate Ligament (ACL) and Posterior Cruciate Ligament (PCL) repair or reconstruction (PCL at US sites only, Biocomposite screw PCL only).

To assess safety, device-related adverse events will be reported and evaluated over the course of the study. To evaluate effectiveness, patient reported outcomes will be collected at 3 months postoperative, 6 months postoperative, and one year postoperative using the Visual Analogue Scale (VAS) for measuring pain in the affected knee and the Knee Injury and Osteoarthritis Outcome Score (KOOS) as well as Range of Motion (ROM, optional) for measuring knee functionality.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires surgery using the Arthrex PEEK Interference Screw for ACL or PCL (PCL at US sites only) repair or reconstruction or the Arthrex Biocomposite Interference Screw for PCL (PCL at US sites only) repair or reconstruction.
* Subject is 18 years of age or over.
* Subject is not considered a vulnerable subject (i.e. child, pregnant, nursing, prisoner, or ward of the state).
* Subject signed informed consent and is willing and able to comply with all study requirements.

Exclusion Criteria:

* Current bilateral injury of the ACL or PCL.
* Injury of the ACL and PCL in the same knee.
* Insufficient quantity or quality of bone.
* Blood supply limitations and previous infections which may retard healing.
* Foreign-body sensitivity.
* Any active infection or blood supply limitations.
* Conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period.
* Subjects that are skeletally immature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 subjects, male and female, at least 18 years of age, will be enrolled for the study. Subjects will be recruited from the surgeon's patient population or referrals from other physicians. The enrollment period is estimated to be 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
To assess change in Visual Analogue Scale (VAS) | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported pain scale 0-10 point scale (0 min, 10 max)
To assess change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported outcome assessment. The interval score ranges from 0 to 100, (where 0 represents total knee disability and 100 represents perfect knee health)
To assess change in Range of Motion (ROM) | preoperatively, 3 months, 6 months and 12 months post operative
  Measuring knee functionality. (Flexion 0 to 130 degrees Extension 120 to 0 degrees

CONTACTS AND LOCATIONS:
Locations (2):
- Anderson Sports Medicine, Bingham Farms, Michigan, United States
- Sportklinik Ravensburg, Ravensburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided